CLINICAL TRIAL: NCT02830529
Title: Mindfulness Attitude to Deliver Dietary Approach to Stop Hypertension
Acronym: MADDASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, KATHY WRIGHT, KL2 Scholar, Postdoc, Case Western Reserve University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: PNR015326A
Record Dates: First submitted 2016-07-05; First posted 2016-07-13 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Prehypertension
Keywords: Mindfulness; African American; fMRI
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MAD DASH (Experimental): Mindfulness based stress reduction and diet education delivered in 8 sessions lasting 2.5 hours each. Mindfulness conducted by a certified trainer. Participants were given homework and meditation CD. Dietitian delivered diet education and conducted interactive food demonstrations. Participants were given option complete weekly diet diary for the dietitian to provide feedback.
  Interventions: Behavioral: MAD DASH; Behavioral: DASH diet education
- DASH diet education (Experimental): Dietary approaches to stop hypertension sessions were delivered by a registered dietitian in 8 sessions lasting 1 hour each. Dietitian delivered diet education and conducted interactive food demonstrations. Participants were given option complete weekly diet diary for the dietitian to provide feedback.
  Interventions: Behavioral: DASH diet education
- Usual Care-DASH Pamphlet Only (No Intervention): Dietary approaches to stop hypertension pamphlet was mailed to each participant. They continued receiving usual care from their health care provider.

INTERVENTIONS:
Behavioral: MAD DASH — Participants were taught mindfulness meditation including body scan, loving kindness meditation and breathing exercises. The diet education component included lecture on reading labels, low cost healthy meal preparation, and dietary consultation regarding personal strengths and self-identified areas of improvement.
  Arms: MAD DASH
Behavioral: DASH diet education — The diet education component included lecture on reading labels, low cost healthy meal preparation, and dietary consultation regarding personal strengths and self-identified areas of improvement.
  Arms: DASH diet education; MAD DASH

SUMMARY:
African Americans with prehypertension have a 35% greater risk of progressing to hypertension than whites. Dietary Approaches to Stop Hypertension (DASH) is a gold standard intervention for hypertension self-management. However, the barriers to self-management of hypertension reported by AAs include stress, including perceived stress related to racism/discrimination; perceived lack of control over getting hypertension in the future; limited social support; and low motivation to change behaviors. Activating the emotional and task areas of the brain are hypothesized to improve self-management behaviors. The purpose of this study is to test the effects of a promising new self-management intervention for AAs, a Mindfulness Attitude to Deliver the Dietary Approach to Stop Hypertension (MAD DASH) that departs from conventional interventions to address prehypertension by combining two self-management interventions (Mindfulness and DASH) in a group setting. Teaching mindfulness; a form of meditation and the DASH diet to participants is expected to result in a reduction in blood pressure as compared to usual care or DASH diet education alone.

DETAILED DESCRIPTION:
Hypertension (HTN), known as the "silent killer" affects 1 in 3 adults in the United States at a cost of $50 billion annually and disproportionately affects African Americans (AA).

A significant proportion of the AA population is living with blood pressures consistent with the clinical criteria for prehypertension or hypertension and many are untreated and undiagnosed. AAs with prehypertension have a 35% greater risk of progressing to hypertension than whites. Salt sensitivity, chronic stress and stress related to racism/discrimination, self-efficacy, motivation, and activation are among the factors associated with pre-HTN in AAs. The prevention of the progression from prehypertension to hypertension through sodium reduction, stress management, and physical activity are a part of the evidence based treatment, but the efficacy of self-management interventions for pre-HTN in AAs is lacking.

The Dietary Approach to Stop Hypertension (DASH) is the gold standard for the prevention and treatment of hypertension yet in many studies, it was reported that AAs were less likely to adhere to the DASH intervention as compared to whites. The barriers to self-management reported by AAs include stress, including perceived stress related to racism/discrimination; perceived lack of control over getting hypertension in the future; limited social support; and low motivation to change behaviors. AAs who perceive stress as the cause of their hypertension are less likely to engage in self-management behaviors. If the brain is in a prolonged state of stress, then the hypothalamic-pituitary-adrenocortical (HPA) activity is compromised leading to allostatic load (wear and tear of chronic stress on the body) increased accumulation of abdominal fat, atrophy of nerve cells in the hippocampus, and hypertension. The interventions used in large hypertension trials do not adequately address chronic stress and effects of racism/discrimination and cognitive mediators (self-efficacy, motivation, activation, decision making, and health information) that hinder the practice of self-management behaviors in AAs. In addition, none of these DASH intervention studies in AAs have included mindfulness, a strategy that has been widely applied across clinical populations to manage obesity, BP, and depression and to motivate patients on a brain level, not just the task level.

Self-management interventions that activate relevant areas of the brain are needed to optimize the adaption of health behaviors. There are two distinctively anti-correlated networks in the brain: analytic brain processing and emotional brain processing that influence self-management behaviors. The analytic brain processing center, located in the prefrontal and parietal areas of the brain is activated during attention demanding tasks (skills, knowledge, and self-monitoring). In contrast, the emotional brain processing center located in the posterior cingulate and medial prefrontal cortices is activated during wakeful rest (emotion management, social cognition, and self-awareness). As the activation of the analytic brain processing center increases, the emotional brain processing center decreases. Thus, a more comprehensive approach that engages both analytic brain processing and emotional brain processing is hypothesized to help AAs to improve motivation, activation and self-efficacy, and garner the necessary social support to succeed in the management of prehypertension. The investigators will test the effects of a promising new self-management intervention for AAs, a Mindfulness Attitude to Deliver the Dietary Approach to Stop Hypertension (MAD DASH) that departs from conventional interventions to address prehypertension by combining two self-management interventions (Mindfulness and DASH) in a group setting.

2) Purpose, specific aims and/or hypotheses

The purpose of this is to gather pilot data to inform a future study using the following aims:

1. Determine whether there are differences in sodium intake, blood pressure (BP), and health related quality of quality of life (HRQoL), among those who receive the analytic component (DASH diet education only), emotional component (MAD-DASH mindfulness plus DASH diet education) compared to those receiving usual care (DASH pamphlet).
2. Examine whether patient activation, motivation, decision-making, self-efficacy, and health information mediate the relationship between the MAD DASH mindfulness intervention and self-management behaviors (diet, self-monitoring, and physical activity).
3. Determine if social support, demographics (gender), and allostatic load moderate the proximal (diet, physical activity) or distal (BP, sodium, and HRQoL) outcomes.
4. Explore differences in brain activation (fMRI) cortical networks, and HPA Axis/stress function (cortisol) among MAD DASH intervention, DASH education only intervention, and usual care.

   3) Background and significance The investigators hypothesize that the MAD DASH intervention will improve the participant's neural brain processing through diet education and self-monitoring and the emotional brain processing level through meditation, deep breathing, and monitoring emotions to promote prehypertension self-management behaviors (diet, self-monitoring, managing emotions, and physical activity). The investigators further hypothesize that these behaviors will lead to a reduction in blood pressure mediated through the HPA axis functioning and stress response (systematic inflammatory effects), cognitive mediators (self-efficacy, decision-making, motivation, health information, and activation), and contextual factors (social support, demographics, allostatic load) to modify the effects of interventions on proximal (increased fruits and vegetables, decreased sodium intake, increased physical activity) and distal (BP, sodium, HRQoL, cost) outcomes. These mechanisms are hypothesized to lead to performance of self-management behaviors, which in turn are expected to lead to subsequent reductions in sodium intake, BP, and improved HRQoL The MAD DASH intervention is likely to improve health behaviors due to integration Mindfulness practice is a non-judgmental self-awareness of emotions, sensations, and cognitions. Mindfulness is believed to affect self-management through self-regulation of responses, acceptance of emotions (e.g., stress, anxiety, and depression), and self-control of emotions---that interfere with the person's ability to practice health behavior management. Improvements in HRQoL are also associated with mindfulness practices. The MAD DASH eight-session intervention will include body scan exercise (lying down or sitting with eyes closed to deliberately focus on sensations within the body), sitting meditation, and yoga exercises along with self-management education (self-monitoring of sodium intake, physical activity) to incorporate strategies to reduce sodium intake, manage emotions, and increase physical activity. There may no direct benefit to subjects, however participation may provide data which will provide insight into ways African Americans can reduce their blood pressure and improve their overall health. Understanding both the biological and psychosocial factors contributing to blood pressure control in African American adults is timely as the population is expected to grow over 9.9 million by 2050 and substantial disparities in health outcomes exist in this population. Findings from this study have the potential to elucidate factors contributing to these disparities in health outcomes in African Americans by better characterization of the neurobiological mechanisms for self-management of prehypertension.

ELIGIBILITY:
Inclusion Criteria:

* African American men or women who:

  * are aged 21 and older,
  * resting systolic (SBP) 120-160 and/or diastolic (DBP) 80-100 mm Hg

Exclusion Criteria:

* diagnosis of hypertension,
* currently taking antihypertensive medication,
* used of glucocorticoids six months prior to inclusion in study,
* adrenal insufficiency,
* expect to move out of the area within six months,
* score less than 20 on the Montreal Cognitive Assessment,
* actively in counseling or regularly (at least three times per week) practice yoga or meditation,
* heart pacemaker, heart defibrillator, metal in the eye, and some types of metal elsewhere within the body such as certain surgical clips for aneurysms in the head, heart valve prostheses, electrodes, and some other implanted devices (for fMRI only), or
* pregnant.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure. | Baseline, 3 months and 9 months.
  Investigators used the JNC-8 criteria for HTN (at or above 140/90 for people under age 60 and 150/90 for persons age 60 and older)

SECONDARY OUTCOMES:
Change in nutrition intake is being changed using the Nutrient Data Systems to assess overall nutrition intake from baseline to 9 months. | 24 hour dietary recall at baseline, 3 months and 9 months.
  Diet recall obtained by the dietician to measure sodium, carbohydrates, sugar, fiber, fruits, and daily caloric intake
Change in physical activity from baseline to 9 months is measured using accelerometry data. | Baseline, 3 months and 9 months
  Accelerometers were programmed and initialized to collect activity counts at one epoch setting and analyzed using ActiLife software.
Change in quality of life from baseline to 9 months was measured using the Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29). | Baseline, 3 months and 9 months
  The PROMIS has 6 subscales for physical function, anxiety, depression, fatigue, social role, and pain.
Change in neuroprocessing from baseline to 3 months will be obtained using functional magnetic resonance imaging | Baseline and 3 months.
  Participants attended a one hour scanner session, which will include collection of a high resolution anatomical image (MPRage) that will allow assessment of gray and while matter density associated with effective self-management as a subsidiary exploratory aim. Participants will then undergo 4 functional runs, each 10 minutes long, which will assess task positive network and the default mode network.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy D Wright, PhD,RN, Principal Investigator — Case Western Reserve University

IPD SHARING:
Plan to Share IPD: Undecided
Yes

REFERENCES:
- [Background] Selassie A, Wagner CS, Laken ML, Ferguson ML, Ferdinand KC, Egan BM. Progression is accelerated from prehypertension to hypertension in blacks. Hypertension. 2011 Oct;58(4):579-87. doi: 10.1161/HYPERTENSIONAHA.111.177410. Epub 2011 Sep 12. PMID 21911708
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Background] Fryar CD, Hirsch R, Eberhardt MS, Yoon SS, Wright JD. Hypertension, high serum total cholesterol, and diabetes: racial and ethnic prevalence differences in U.S. adults, 1999-2006. NCHS Data Brief. 2010 Apr;(36):1-8. PMID 20423605
- [Background] Richardson SI, Freedman BI, Ellison DH, Rodriguez CJ. Salt sensitivity: a review with a focus on non-Hispanic blacks and Hispanics. J Am Soc Hypertens. 2013 Mar-Apr;7(2):170-9. doi: 10.1016/j.jash.2013.01.003. Epub 2013 Feb 19. PMID 23428408
- [Background] Pal GK, Chandrasekaran A, Hariharan AP, Dutta TK, Pal P, Nanda N, Venugopal L. Body mass index contributes to sympathovagal imbalance in prehypertensives. BMC Cardiovasc Disord. 2012 Jul 19;12:54. doi: 10.1186/1471-2261-12-54. PMID 22812583
- [Background] Dolezsar CM, McGrath JJ, Herzig AJM, Miller SB. Perceived racial discrimination and hypertension: a comprehensive systematic review. Health Psychol. 2014 Jan;33(1):20-34. doi: 10.1037/a0033718. PMID 24417692
- [Background] Bavikati VV, Sperling LS, Salmon RD, Faircloth GC, Gordon TL, Franklin BA, Gordon NF. Effect of comprehensive therapeutic lifestyle changes on prehypertension. Am J Cardiol. 2008 Dec 15;102(12):1677-80. doi: 10.1016/j.amjcard.2008.08.034. Epub 2008 Oct 23. PMID 19064023
- [Background] Appel LJ, Champagne CM, Harsha DW, Cooper LS, Obarzanek E, Elmer PJ, Stevens VJ, Vollmer WM, Lin PH, Svetkey LP, Stedman SW, Young DR; Writing Group of the PREMIER Collaborative Research Group. Effects of comprehensive lifestyle modification on blood pressure control: main results of the PREMIER clinical trial. JAMA. 2003 Apr 23-30;289(16):2083-93. doi: 10.1001/jama.289.16.2083. PMID 12709466
- [Background] Epstein DE, Sherwood A, Smith PJ, Craighead L, Caccia C, Lin PH, Babyak MA, Johnson JJ, Hinderliter A, Blumenthal JA. Determinants and consequences of adherence to the dietary approaches to stop hypertension diet in African-American and white adults with high blood pressure: results from the ENCORE trial. J Acad Nutr Diet. 2012 Nov;112(11):1763-73. doi: 10.1016/j.jand.2012.07.007. Epub 2012 Sep 19. PMID 23000025
- [Background] Pickett S, Allen W, Franklin M, Peters RM. Illness beliefs in African Americans with hypertension. West J Nurs Res. 2014 Feb;36(2):152-70. doi: 10.1177/0193945913491837. Epub 2013 Jun 13. PMID 23765710
- [Background] Flynn SJ, Ameling JM, Hill-Briggs F, Wolff JL, Bone LR, Levine DM, Roter DL, Lewis-Boyer L, Fisher AR, Purnell L, Ephraim PL, Barbers J, Fitzpatrick SL, Albert MC, Cooper LA, Fagan PJ, Martin D, Ramamurthi HC, Boulware LE. Facilitators and barriers to hypertension self-management in urban African Americans: perspectives of patients and family members. Patient Prefer Adherence. 2013 Aug 6;7:741-9. doi: 10.2147/PPA.S46517. eCollection 2013. PMID 23966772
- [Background] Kressin NR, Orner MB, Manze M, Glickman ME, Berlowitz D. Understanding contributors to racial disparities in blood pressure control. Circ Cardiovasc Qual Outcomes. 2010 Mar;3(2):173-80. doi: 10.1161/CIRCOUTCOMES.109.860841. Epub 2010 Jan 19. PMID 20233981
- [Background] McEwen BS, Gianaros PJ. Central role of the brain in stress and adaptation: links to socioeconomic status, health, and disease. Ann N Y Acad Sci. 2010 Feb;1186:190-222. doi: 10.1111/j.1749-6632.2009.05331.x. PMID 20201874
- [Background] Mainous AG 3rd, Everett CJ, Liszka H, King DE, Egan BM. Prehypertension and mortality in a nationally representative cohort. Am J Cardiol. 2004 Dec 15;94(12):1496-500. doi: 10.1016/j.amjcard.2004.08.026. PMID 15589003
- [Background] Kwan MW, Wong MC, Wang HH, Liu KQ, Lee CL, Yan BP, Yu CM, Griffiths SM. Compliance with the Dietary Approaches to Stop Hypertension (DASH) diet: a systematic review. PLoS One. 2013 Oct 30;8(10):e78412. doi: 10.1371/journal.pone.0078412. eCollection 2013. PMID 24205227
- [Background] Palta P, Page G, Piferi RL, Gill JM, Hayat MJ, Connolly AB, Szanton SL. Evaluation of a mindfulness-based intervention program to decrease blood pressure in low-income African-American older adults. J Urban Health. 2012 Apr;89(2):308-16. doi: 10.1007/s11524-011-9654-6. PMID 22302233
- [Background] Fjorback LO, Arendt M, Ornbol E, Fink P, Walach H. Mindfulness-based stress reduction and mindfulness-based cognitive therapy: a systematic review of randomized controlled trials. Acta Psychiatr Scand. 2011 Aug;124(2):102-19. doi: 10.1111/j.1600-0447.2011.01704.x. Epub 2011 Apr 28. PMID 21534932
- [Background] Hamilton JP, Furman DJ, Chang C, Thomason ME, Dennis E, Gotlib IH. Default-mode and task-positive network activity in major depressive disorder: implications for adaptive and maladaptive rumination. Biol Psychiatry. 2011 Aug 15;70(4):327-33. doi: 10.1016/j.biopsych.2011.02.003. Epub 2011 Apr 3. PMID 21459364
- [Background] Hughes JW, Fresco DM, Myerscough R, van Dulmen MH, Carlson LE, Josephson R. Randomized controlled trial of mindfulness-based stress reduction for prehypertension. Psychosom Med. 2013 Oct;75(8):721-8. doi: 10.1097/PSY.0b013e3182a3e4e5. PMID 24127622
- [Background] Friese M, Messner C, Schaffner Y. Mindfulness meditation counteracts self-control depletion. Conscious Cogn. 2012 Jun;21(2):1016-22. doi: 10.1016/j.concog.2012.01.008. Epub 2012 Feb 5. PMID 22309814
- [Derived] Wright KD, Jack AI, Friedman JP, Jones LM, Sattar A, Fresco DM, Moore SM. Neural Processing and Perceived Discrimination Stress in African Americans. Nurs Res. 2020 Sep/Oct;69(5):331-338. doi: 10.1097/NNR.0000000000000441. PMID 32496401
- [Derived] Moore SM, Musil CM, Alder ML, Pignatiello G, Higgins P, Webel A, Wright KD. Building a Research Data Repository for Chronic Condition Self-Management Using Harmonized Data. Nurs Res. 2020 Jul/Aug;69(4):254-263. doi: 10.1097/NNR.0000000000000435. PMID 32205788
- [Derived] Moore SM, Musil CM, Jack AI, Alder ML, Fresco DM, Webel A, Wright KD, Sattar A, Higgins P. Characterization of Brain Signatures to Add Precision to Self-Management Health Information Interventions. Nurs Res. 2019 Mar/Apr;68(2):127-134. doi: 10.1097/NNR.0000000000000331. PMID 30540702